CLINICAL TRIAL: NCT07151781
Title: Technology Supported Mindfulness for Prenatal Depression and Mental Health-related Quality of Life: Research Protocol for Randomized Controlled Trial in a Resource-Limited Environment
Brief Title: Technology Supported Mindfulness for Prenatal Depression and Mental Health-related Quality of Life in a Resource-Limited Environment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bekelu Teka Worku (Other)
Collaborators: Jimma University (Other)
Responsible Party: Sponsor-Investigator, Bekelu Teka Worku, Principal Investigator, Jimma University
Organization: Jimma University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JUIH/IRB/425/24
Record Dates: First submitted 2025-08-19; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Prenatal Depression; Mental Health Related Quality of Life; Maternal Postpartum Depression; Paternal Postpartum Depression
Keywords: mHealth; mindfulness; prenatal depression; randomized controlled trial; health technology; RCT

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial (RCT) with a 1:1 allocation ratio will be used to compare a video-guided mindfulness intervention group with a standard care control group.
  Study participants will be recruited at the community level. Pregnant women will be identified and registered by a team called "Gaachana", a local volunteer group working under the supervision of Health Extension Workers (HEWs). Screening for PND will be conducted using the Edinburgh Postnatal Depression Scale (EPDS) by trained data collectors until the required sample size is achieved. Eligible participants will be randomly assigned to either the intervention or control group.
Who Masked: Care Provider
Masking Description: Data collectors Participants in the control arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): The intervention arm will receive a video-guided mindfulness practice consisting of audio recordings (in two local languages: Afan Oromo and Amharic) combined with familiar natural environment visuals. The exercise instruction consists of three core mindfulness practices: (i) Focus the Mind: to cultivate present-moment attention and reduce cognitive rumination; (ii) Breath Awareness: to anchor attention and promote relaxation; and (iii) Basic Body Scan: to encourage non-judgmental awareness of bodily sensations to enhance their mind-body connection.
  The intervention will be delivered face-to-face at the health centers using a smartphone-based video. The intervention is planned to be delivered regularly according to a standardized schedule for each of the women individually. Each session of the exercise can last for about 21-23 minutes. Hired Midwifery Nurses at each of the health centers will support the woman to start the exercise and follow her till the end of the sessions daily.
  Interventions: Other: Video-guided Mindfulness Exercise
- Control group (No Intervention): The control group will continue with the routine maternal and other standard health care services as provided by the health centers in accordance with national maternal health guidelines. In Ethiopia, according to the National Antenatal Care Guideline 2022, each woman must visit the health facility for eight contacts. They are expected to screened for potentially recurring obstetric complications such as recurrent pregnancy loss, preterm labor, pre-eclampsia/eclampsia, gestational diabetes, congenital anomaly, puerperal psychosis, obstetric and gynecologic surgery, immunologic disorders, medical and mental health disorders, infectious diseases, physical disability and developmental disorders, nutritional history, social and personal history, current medication, and intimate partner violence. They receive counselling on the risk of pregnancy, contraception, micronutrient supplementation, weight gain monitoring, counselling on the increased risk to the fetus, and other related services.

INTERVENTIONS:
Other: Video-guided Mindfulness Exercise — Mindfulness interventions are emerging as effective, low-risk approaches to managing depression and enhancing emotional and maternal well-being in pregnant women. Rooted in ancient meditative practices that originated from Buddhist religion and traditions and adapted for clinical use, mindfulness intervention cultivates present-moment awareness and nonjudgmental acceptance of thoughts, emotions, and bodily sensations. Mostly, mindfulness interventions include elements such as mindful breathing and body scanning and have shown effectiveness in reducing depressive symptoms and enhancing emotional regulation. It is the ability to maintain attention to an immediate experience with a sense of adopting an open and accepting attitude toward that experience. However, further research is important to evaluate its effectiveness across diverse sociodemographic and socioeconomic settings.
  Arms: Intervention arm

SUMMARY:
The goal of this clinical trial is to learn if a video-guided mindfulness intervention can improve prenatal depression symptoms, improve mental health-related quality of life, reduce the risk of maternal postpartum depression and paternal postpartum depression, and improve neonatal birth outcomes in a resource-constrained setting. This clinical trial will be conducted in pregnant women. The main questions it aims to answer are:

* Can video-guided mindfulness intervention be effective for prenatal depression treatment as compared to routine care?
* Is there a dose-response relationship between the length of a video-guided mindfulness intervention and a reduction in prenatal depression symptoms?
* Does a video-guided mindfulness intervention improve mental health-related quality of life more effectively than routine care?
* What is the impact of intervention duration on the effectiveness of a video-guided mindfulness intervention for improving mental health-related quality of life?
* Can a video-guided mindfulness intervention during pregnancy lead to improved neonatal birth outcomes compared to standard care?
* Can a video-guided mindfulness intervention during pregnancy reduce the risk of developing prenatal depression compared to routine care?
* Can the treatment of maternal prenatal depression through a video-guided mindfulness intervention reduce the risk of paternal postpartum depression? Researchers will compare the intervention group with a group of pregnant women who screen positive for prenatal depression but continue to receive only routine antenatal care, in order to evaluate differences in prenatal depression symptoms, improvements in mental health-related quality of life, reductions in the risk of maternal and paternal postpartum depression, and improvements in neonatal birth outcomes.

Participants (the intervention group) will receive a video-guided mindfulness intervention that they will listen to for eight weeks at their nearest health center three times a week.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who lived in Jimma City for at least six months
* Women with a gestational age between 12 and 28 weeks,
* Women who scored EPDS ≥ 13,
* Willing to participate for eight consecutive weeks,
* Able to attend the health center three times per week and gave consent to be followed up by study supervisors and data collectors

Exclusion Criteria:

* Having been diagnosed with mental health disorders or eating disorders,
* Active substance use,
* EPDS item 10 score ≥1 or total EPDS score >19,
* Currently receiving pharmacological or psychotherapeutic treatment,
* Regularly practice meditation,
* Severely ill,
* Has active pregnancy-related complications that could interfere with attending the mindfulness exercise, or neurological conditions such as epilepsy or seizures

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Prenatal Depression Symptoms | The primary outcome will be assessed immediately after the intervention is done; after eight weeks of the initiation of the intervention.
  The symptoms of prenatal depression will be measured using the Edinburgh Postnatal Depression Scale. The EPDS is a widely validated 10-item self-report questionnaire designed to screen depressive symptoms primarily in the postnatal period and later extended for prenatal period depression symptoms. The study participants will be asked to report their relevant rating scale out of the available four response options with the EPDS. They will be asked about their experience of the symptoms over the past seven days. The higher score, which is three, indicates greater levels of depressive symptoms, and a zero score shows the absence of the symptoms. The maximum total score in EPDS is 30, where a cut-off score of ≥13 in clinical and research settings is used to indicate positive screened for PND.

SECONDARY OUTCOMES:
Better Mental Health Related Quality of Life | Mental Health Related Quality of Life will be evaluated immediately after intervention (After eight weeks).
  The Mental Health Related Quality of Life (MHRQoL) will be assessed using the Mental Health Quality of Life-7 Dimensions (MHQoL-7D) questionnaire. The MHQoL-7D helps to evaluate seven key dimensions of mental health and well-being. The seven dimensions include "self-image, independence, mood, relationships, daily activities, physical health, and future outlook" of the individuals. This tool contains seven questions with a five-point Likert scale and measures feelings of the individual over the day. The score in MHQoL-7D ranges from a minimum of 0 to a maximum of 21, with the lower score indicating poor MHRQoL.

OTHER OUTCOMES:
Symptoms of maternal postpartum depression | Symptoms of maternal postpartum depression will be measured at the ninth week from initiation of intervention.
  The symptoms of maternal postpartum depression will be measured using the Edinburgh Postnatal Depression Scale. The EPDS is a widely validated 10-item self-report questionnaire designed to screen depressive symptoms primarily in the postnatal period and later extended for prenatal period depression symptoms. The study participants will be asked to report their relevant rating scale out of the available four response options with the EPDS. They will be asked about their experience of the symptoms over the past seven days. The higher score, which is three, indicates greater levels of depressive symptoms, and a zero score shows the absence of the symptoms. The maximum total score in EPDS is 30, where a cut-off score of ≥13 in clinical and research settings is used to indicate positive screened for postpartum depression.
Symptoms of paternal postpartum depression | Symptoms of paternal postpartum depression will be measured at the ninth week from initiation of intervention.
  The symptoms of paternal postpartum depression will be measured using the Edinburgh Postnatal Depression Scale. The EPDS is a widely validated 10-item self-report questionnaire designed to screen depressive symptoms primarily in the postnatal period and later extended for prenatal period depression symptoms. The study participants will be asked to report their relevant rating scale out of the available four response options with the EPDS. They will be asked about their experience of the symptoms over the past seven days. The higher score, which is three, indicates greater levels of depressive symptoms, and a zero score shows the absence of the symptoms. The maximum total score in EPDS is 30, where a cut-off score of ≥13 in clinical and research settings is used to indicate positive screened for postpartum depression.
Neonatal birth outcome | Neonatal birth outcome will be assessed at the ninth week from initiation of intervention.
  Neonatal birth outcome will be assessed using a developed tool.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Bonnechere, PhD, Principal Investigator — Hasselt University; Misra Abdulahi, PhD, Principal Investigator — Jimma University; Demissew Amenu Sori, PhD, Principal Investigator — Jimma University
Locations (1):
- Jimma City in the Southwestern part of Ethiopia, 353 km away from the capital city, Addis Ababa., Jimma, Ethiopia

IPD SHARING:
Plan to Share IPD: Undecided
The data will be published in aggregate form without any information that could identify individual participants. If additional information is requested by other researchers, I may share the data in an anonymized format, and only when its use serves the advancement of scientific knowledge and aligns with the best interests of the study participants.

REFERENCES:
- [Background] Worku BT, Abdulahi M, Amenu D, Bonnechere B. Effect of technology-supported mindfulness-based interventions for maternal depression: a systematic review and meta-analysis with implementation perspectives for resource-limited settings. BMC Pregnancy Childbirth. 2025 Feb 13;25(1):155. doi: 10.1186/s12884-025-07286-9. PMID 39948517
- [Background] 1. Molenaar NM, Kamperman AM, Boyce P, Bergink V. Guidelines on treatment of perinatal depression with antidepressants: an international review. Australian & New Zealand Journal of Psychiatry. 2018;52(4):320-7. 2. Leng LL, Yin XC, Ng SM. Mindfulness-based intervention for clinical and subthreshold perinatal depression and anxiety: a systematic review and meta-analysis of randomized controlled trial. Comprehensive Psychiatry. 2023;122:152375. 3. Min W, Jiang C, Li Z, Wang Z. The effect of mindfulness-based interventions during pregnancy on postpartum mental health: a meta-analysis. J Affect Disord. 2023;331:452-60. 22. Marlatt GA. Buddhist philosophy and the treatment of addictive behavior. Cogn Behav Pract. 2002;9(1):44-50. 4. Kabat-Zinn J. Mindfulness-based stress reduction (MBSR). Constructivism in the human sciences. 2003;8(2):73.